CLINICAL TRIAL: NCT04823962
Title: Effect of Topical rhGM-CSF on the Healing of Venous Leg Ulcers: a Randomized, Placebo-controlled, Double-blind, Clinical Phase II Study
Brief Title: Effect of rhGM-CSF on the Healing of Venous Leg Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reponex Pharmaceuticals A/S (Industry)
Responsible Party: Principal Investigator, Torsten Bjørn, Prinicipal Investigator, MD, Reponex Pharmaceuticals A/S
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Repogel-01
Record Dates: First submitted 2021-03-06; First posted 2021-04-01 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — regramostim; Hydrogels; molgramostim; Standard of Care

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled and double-blind, phase II clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GM-CSF (Experimental): rhGM-CSF (molgramostim) + hydrogel
  Interventions: Drug: rhGM-CSF + hydrogel; Other: Standard care
- Placebo (Placebo Comparator): Hydrogel
  Interventions: Drug: Placebo hydrogel; Other: Standard care

INTERVENTIONS:
Drug: rhGM-CSF + hydrogel — The active substance: molgramostim (rhGM-CSF)
  Other Names: Repogel; Molgramostim
  Arms: GM-CSF
Drug: Placebo hydrogel — Placebo hydrogel
  Arms: Placebo
Other: Standard care — Compression therapy and neutral dressings

SUMMARY:
The objective of this study is to examine whether local administration of the growth factor rhGM-CSF incorporated into a hydrogel, can accelerate wound healing when applied to venous leg ulcers, and whether this is safe.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged aged 18 years or older
2. Patients with at least one difficult-to-heal venous leg ulcer on standard care (diagnosed by clinical evaluation) localized between the knee and ankle, including the perimalleolar area.
3. Venous insufficiency confirmed by a venous Doppler/duplex ultrasound scan. A previous scan before randomization can be used. If there is no previous adequate scanning, a new scanning has to be performed before randomization.
4. Ulcer size 2-75 cm2 at randomization day (D0), the upper limit being defined as the largest ulcer in size that fits the area selection criteria
5. Ulcer duration ≥2 months and ≤3 years
6. Negative p-HCG for women of childbearing potential
7. Patient able to understand Danish
8. Patient able to comply with the protocol
9. Patient fully informed about the study and having given written informed consent

Exclusion Criteria:

1. Characteristics of the index ulcer:

   1. Exposed bone, tendon, ligament, cartilage, joint or muscle
   2. Cellulitis or clinical ulcer infection at the screening day D-4, or the day of randomization, D0.
   3. Ulcers adjacent to the index ulcer that could interfere with the index ulcer, as judged by investigator
2. Patients that are unsuitable for the compression therapy used in the study
3. Known allergy towards GM-CSF, excipients or any other substances or remedies used in the trial.
4. Vascularization: Ankle-brachial index ≤0.7
5. Active or history of following diseases:

   1. Cancer (past history of well-treated cancer is however accepted after a control period of more than two years).
   2. Following autoimmune diseases: rheumatoid arthritis, autoimmune thrombocytopenia, thyroiditis, psoriasis, nephritis or multiple sclerosis.
   3. Lower extremity deep venous thrombosis within the last 3 months
6. Any of following active diseases:

   1. Serious heart disease, including unstable angina pectoris, a major cardiac event such as myocardial infarction, congestive heart failure NYHA class III-IV within 3 months before the study
   2. Neutrophilic dermatoses (e.g. pyoderma gangrenosum and Sweet's syndrome)
   3. Severe renal-, hepatic or pulmonary insufficiency or severely dysregulated diabetes, as judged by investigator
   4. Myeloproliferative diseases and hematologic diseases (e.g. myelodysplastic syndrome and leukemia). Anemia due to chronic infection or due to deficiency of iron, B12 or folic acid is accepted if Hb >5 mmol/L).
   5. Significant dementia
7. Biochemistry with clinically significant abnormalities that could preclude study participation as judged by the investigator, such as:

   1. eGFR <20 mL/min/1.73 m2
   2. Hb <5 mmol/L
   3. ALAT >1.5 x upper limit of normal value
   4. Albumin < 20 g/l
8. Prohibited therapy:

   1. Systemic immunosuppressive treatment, immunomodulators, cytotoxic chemotherapy (exception: usage of corticosteroids) on D-4 or D0.
   2. Corticosteroids with a daily dose equivalent to >10 mg of prednisolone per day on D-4 or D0.
   3. Topical corticosteroids in the index ulcer bed or within 1 cm of the ulcer edge on D-4 or D0.
   4. Biologics within 3 months of D-4 (anti-VEGF treatment in the eye in e.g. diabetics is however allowed).
9. Weight <50 kg or BMI >50
10. Participation in another clinical trial
11. Planned surgery or hospitalization during trial
12. Pregnant or lactating woman. Positive pregnancy test during run-in.
13. Failure to agree to using an adequate method of contraception (having a failure rate of < 1% per year) throughout the study period for heterosexually active males and females of childbearing potential, or disagreement to remain abstinent (refrain from heterosexual intercourse). A woman is considered to be of childbearing potential if she is post-menarche and:

    1. Has not reached a postmenopausal state (≥60 years of age and amenorrhea for at least ≥12 months with no identified cause other than menopause, and has not undergone surgical sterilization: removal of ovaries and/or uterus) - OR
    2. No menses for over a year and confirmed by follicle-stimulating hormone (FSH) levels elevated into the postmenopausal range Examples of contraceptive methods with a failure rate of <1% per year includes bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives, hormone-releasing intrauterine devices and copper intrauterine devices. Male participants must be abstinent or use a condom during the trial period.
14. Blood or sperm donation during trial
15. Patient has previously been randomized in this study (rescreening is accepted otherwise)
16. Judgment by the investigator that the patient is not suited for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching a 40% ulcer area reduction, or more, 4 weeks after initiation of the study drug treatment/placebo | 4 weeks after initiation of the study drug treatment/placebo
  Ulcer size (area in cm2) will be assessed on the randomization day (Day 0; initiation of the study drug treatment/placebo) and at the end of the study drug/placebo treatment (D28+1)

SECONDARY OUTCOMES:
Absolute change of the ulcer area | 4 and 8 weeks after randomization
  The ulcer size is compared in terms of change in cm2 from the randomization day
Percentage change of the ulcer area | 4 and 8 weeks after randomization
  The ulcer size is compared in terms of percentage change from the randomization day
Complete ulcer healing | 4 and 8 weeks after randomization
  Number of subjects reaching complete ulcer healing; Full epithelization and no drainage of wound fluid or dressing requirements
Time to complete ulcer healing | Through study completion (8 weeks)
  Time to complete ulcer healing in days, with the randomization day as baseline
Clinical improvement of the wound healing process | 4 and 8 weeks after randomization
  Semi-quantitatively measured (major improvement, minor improvement, status quo or worsening)
Assessment of the safety profile | Throughout the trial (8 weeks)
  All clinical and laboratory adverse events will be assessed and recorded.

OTHER OUTCOMES:
Exploratory measurement: Changes in the levels of cytokines and growth factors in the wound fluid | Wound fluid is collected at three time points: Before initiation of the study drug/placebo (Day 0), after two weeks of treatment (Day 14) and at the end of the treatment period (Day 28).
  Changes in the levels of each cytokine and growth factor will be quantified over time
Exploratory measurement: Wound status | Throughout the trial (8 weeks)
  Degree of inflammation, granulation tissue, necrosis/slough, exudation and infection. Semi-quantitatively measured.
Exploratory measurement: Changes in the microbiome (number of viable bacteria) | Before initiation of study drug and after two weeks of treatment
  Assessed by the colony-forming unit (CFU)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa A Burian, MD, Principal Investigator — Department of Dermatology and Copenhagen Wound Healing Center
Locations (1):
- Department of Dermatology and Copenhagen Wound Healing Center, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No